CLINICAL TRIAL: NCT06217224
Title: Evaluation of Prophylactic Photobiomodulation Therapy in Patients With Osteosarcoma Undergoing High Doses of Methotrexate
Brief Title: Evaluation of Prophylactic Photobiomodulation Therapy in Patients With Osteosarcoma
Acronym: PBMT/MTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Heliton Spindola Antunes, Doctor of oncology, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 54417221.3.0000.5274
Record Dates: First submitted 2023-11-21; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Mucositis Oral
Keywords: osteosarcoma; Mucositis Oral; Methotrexate Toxicity; Low-Level Light Therapy
MeSH Terms: conditions — Stomatitis; Osteosarcoma

STUDY DESIGN:
Intervention Model Description: Phase 3, randomized study with patients diagnosed with OS, enrolled at INCA, candidates for the Glato protocol (chemotherapy -doxorubicin, cisplatin, dexamethasone and MTX + surgery). Patients will be randomized through the computerized system to groups 1 or 2.
  Randomization will be performed in permuted blocks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventative photobiomodulation therapy arm only in methotrexate weeks. (Active Comparator): The application of preventive photobiomodulation therapy (PBMT) will be carried out on the day of methotrexate infusion (D1) and until the patient reaches a serum concentration equal to or less than 0.3 mmol/L.
  Interventions: Other: Preventive photobiomodulation Therapy (PBMT)
- Preventive photobiomodulation therapy arm in the weeks of methotrexate, cisplatin and doxorubicin. (Experimental): The application of preventive photobiomodulation therapy will be performed on the days of doxorubicin infusion and cisplatin and on the day after the doxorubicin infusion; on the day of the methotrexate infusion and until the patient reaches a serum concentration equal to or less than 0.3 mmol /L.
  Interventions: Other: Preventive photobiomodulation Therapy (PBMT)

INTERVENTIONS:
Other: Preventive photobiomodulation Therapy (PBMT) — The application of preventive TLBP will be performed with a laser device containing an aluminum phosphide and indium gallium diode (InGaAlP) emitting radiation in the red region of the electromagnetic spectrum (660 nm) with a power of 100mW and a beam area of 0.03 cm2 . An energy of 1J/point and an energy density of 33.3 J/cm2/point were determined, which will be applied punctually, with a distance between the points of 1cm, for 10s per point, totaling 9 points per region.
  Other Names: Preventive Low Power Laser Therapy (TLBP )

SUMMARY:
This study aims to evaluate the photobiomodulation therapy (PBMT) for the prevention of oral mucositis in osteosarcoma patients submitted to high doses of methotrexate, through two different protocols. As a hypothesis, photobiomodulation for the prevention of oral mucositis after cycles of Cisplatin, Doxorubicin and Methotrexate is more effective than just the application of preventive low-power laser after Methotrexate alone.

DETAILED DESCRIPTION:
This is a phase 3, randomized study, with patients diagnosed with osteosarcoma, enrolled at national cancer institute in Brazil (INCA), candidates for the Glato protocol (chemotherapy with doxorubicin, cisplatin, methotrexate and surgery). Patients will be randomly randomized in permuted blocks to groups 1 or 2. After confirming the eligibility criteria, patients will be invited to participate in the research before starting treatment and the TCLE/TALE will be applied in accordance with the Good Clinical Practice Guide and national ethical standards.

After signing the TALE/TCLE, patients will be instructed to perform oral hygiene after all meals, solid or liquid, with fluoridated toothpaste. On the first day of chemotherapy, in addition to the oral hygiene protocol, patients will be instructed to rinse their mouth twice a day with 0.12% chlorhexidine for 7 days. Once hyposalivation is diagnosed, patients will use oral humidifying gel four times a day (brand provided by the institution).

Photobiomodulation therapy

* Preventative photobiomodulation therapy will be performed with the MMO device (São Carlos, São Paulo, Brazil), with an indium gallium aluminum phosphide (InGaAlP) diode with radiation emission in the red region of the electromagnetic spectrum (660 nm) with power of 100mW, with a beam area of 0.03cm². An energy of 1J/point and an energy density of 33.3 J/cm²/point were determined, which will be applied punctually, with a distance between points of 1cm, for 10s per point, totaling 9 points per region .
* The technique will be performed on the first day of methotrexate infusion and until the patient reaches a serum concentration equal to or lower than 0.3 mmol/L; on the days of doxorubicin and cisplatin infusion and the day after; and on the days of infusion of doxorubicin alone in weeks 24 and 28 of the Glato protocol. Photobiomodulation will be performed in all cycles of chemotherapy treatment depending on patient randomization.
* Group 1- Preventive photobiomodulation will be carried out on the day of methotrexate infusion and until the patient reaches a serum concentration equal to or lower than 0.3 mmol/L, from weeks 4, 5, 9, 10, 17, 18, 22, 23 , 26, 27, 30 and 31). On the days of infusion of doxorubicin and cisplatin and doxorubicin isoleted, patients will not receive photobiomodulation therapy.
* Group 2- Preventative photobiomodulation will be carried out on the days of doxorubicin infusion (weeks 1, 6, 14, 19, 24 and 28) and cisplatin (weeks 1, 6, 14 and 19) and on the day after doxorubicin infusion and cisplatin (weeks 1, 6, 14, 19), on the days of infusion of doxorubicin isoleted, weeks 24 and 28, photobiomodulation will be performed only on the first and second day. The technique will also be performed on the day of methotrexate infusion and on subsequent days until the patient reaches a serum concentration equal to or less than 0.3 mmol/L, from weeks 4, 5, 9, 10, 17, 18, 22, 23 , 26, 27, 30 and 31).
* If the patient presents oral mucositis Grade 1, 2, 3 or 4, they will receive treatment with the MMO device (São Carlos, São Paulo, Brazil), with an indium gallium aluminum phosphide diode (InGaAlP) with radiation emission in the red region of the electromagnetic spectrum (660 nm) with a power of 100mW, with a beam area of 0.03cm². An energy of 2J/point and an energy density of 66.6 J/cm²/point were determined, which will be applied punctually, for 20s per point in the area with MO and in healthy areas.
* The regions treated with laser of the oral mucosa will be: right and left buccal mucosa, lower and upper lip, upper and lower labial mucosa, right and left lateral border of the tongue, lingual belly, floor of the mouth and soft palate.
* Assessment of the patient's oral mucosa will be carried out by members of the research project team.

Oral assessment

Patients will be evaluated at the beginning of chemotherapy treatment (D1) and in a second moment between the third and seventh subsequent days (D3 to D7). In weeks 24 and 28, the dental evaluation will be carried out on D1 and between the second and seventh day (D2 to D7). In the weeks when the patient does not attend the hospital, a teleconsultation will be carried out to monitor the symptoms and, if a need for face-to-face evaluation is identified, an appointment will be scheduled.The mucous membranes will be evaluated for color, hydration, integrity, presence of oral mucositis and fungal, bacterial and viral infections.

The assessment of oral mucositis will be established according to the 1979 World Health Organization (WHO) classification and the criteria established by Sonis et al in 1999 (OMAS). The WHO assessment scale is made up of: Grade 0 - no change (Absent); Grade 1 - presence of erythema; Grade 2 - presence of erythema and ulcers, but the patient is able to ingest solids and liquids; Grade 3 - presence of ulcers, but the patient can only ingest a liquid and pasty diet and Grade 4 - presence of ulcers and impossibility of ingesting solids or liquids.

The OMAS scale considers the presence and size of ulcerations/pseudomembranes and erythema. Ulcerations/pseudomembranes will be evaluated according to the following scores: 0 - in the absence of lesions, 1 - in lesions smaller than 1 cm3, 2 - in lesions measuring between 1 and 3 cm3 and 3 - in lesions larger than 3cm3. Erythema will be evaluated according to the following scores: 0 - when absent, 1 - when present but not severe and 2 - when present and severe. A daily calculation will be made of the sum of the weighted average of the ulcerated area and intensity of the erythema (MP=2.5 x [(∑ui : 3 x Nu )+ (∑ei: 2 x Ne) ], where ∑ ui= sum of ulcerated area, Nu= number of ulcerated areas, ∑ei= sum of erythema intensity and Ne= number of areas with erythema A millimeter dental ruler will be used to measure the area.

Patients will be asked about the presence or absence of oral and oropharyngeal pain. Both will be classified according to CTCAE v5.0 into grades 1, 2 and 3, associated with the Visual Analogue Scale, where the value 0 corresponds to no pain and 10, the greatest pain. According to the standards established by the visual analogue scale, values from 0 to 3 correspond to mild pain, from 4 to 6 to moderate pain and from 7 to 10 to severe pain.

The collection of adverse events will only be directed to events of interest to the study, related to toxicities in the oral cavity. It is not expected that there will be collection and analysis of serious adverse events in this study.

Xerostomia will be assessed according to the presence or absence of complaints about this condition on the part of the patient, associated with sialometry according to CTCAE v5.0 in grades 1, 2 and 3, on the first day of each chemotherapy cycle and between the third and seventh day (D3 and D7) of the same week of chemotherapy. In weeks 24 and 28, salivary flow will be assessed on the first day (D1) and between the second and seventh day (D2 to D7).

Unstimulated saliva collection will be performed according to the method described by Davies et al. (2002) The patient will remain seated vertically in a comfortable place. The first saliva sample will be discarded and the rest will be collected in a decontaminated bottle. The collected saliva will be converted into ml/minute and an unstimulated salivary flow of less than 0.1mL/min will be considered hyposalivation. Clinical criteria will also be used to identify xerostomia, such as sublingual salivary lake, salivary thickening and adherence of the wooden spatula to the oral mucosa, associated with the patient's complaint.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled at INCA diagnosed with OS (ICD10-C41), aged 0 to 19 years;
* Patients with indication for Glato chemotherapy protocol, which will use high doses of MTX (HD-MTX (>1 g/m2).
* Patients who, after receiving information and instructions, signed the patient's informed consent/assent form, in accordance with Resolution 466/12 of the National Health Council.

Exclusion Criteria:

- Patients who do not agree with the proposed treatment.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the best photobiomodulation protocol for preventing oral mucositis | Throughout the entire glato protocol.
  To compare the effectiveness of two photobiomodulation protocols for the prevention of oral mucositis in patients with osteosarcoma undergoing high doses of methotrexate.

SECONDARY OUTCOMES:
Incidence of Oral Mucositis | From the first day of infusion of each chemotherapy agent to the third and seventh day of the same week of infusion throughout the entire glato protocol.
  Compare the duration of oral mucositis in patients undergoing preventive photobiomodulation in groups 1 (only in the chemotherapy cycle of methotrexate) and group 2 (in cycles of methotrexate, doxorubicin and cisplatin).
Oral mucositis development time | From the first day of infusion of each chemotherapy agent to the third and seventh day of the same week of infusion throughout the entire glato protocol.
  Evaluate the development time of oral mucositis following the chemotherapy cycle.
Assess salivary flow | From the first day of infusion of each chemotherapy agent to the third and seventh day of the same week of infusion throughout the entire glato protocol.
  Assess salivary flow before starting the first cycle of chemotherapy and in subsequent consultations.
Methotrexate serum levels | From the first day of meotrexate infusion until serum regularization.
  Assess serum methotrexate levels after chemotherapy infusion, until they are regularized, during the study.
Hospital internment | Throughout the entire glato protocol.
  To evaluate the frequency of hospital admissions due to adverse events of interest to the study during chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Heliton S Antunes, Dr., Study Director — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Steliarova-Foucher E, Colombet M, Ries LAG, Moreno F, Dolya A, Bray F, Hesseling P, Shin HY, Stiller CA; IICC-3 contributors. International incidence of childhood cancer, 2001-10: a population-based registry study. Lancet Oncol. 2017 Jun;18(6):719-731. doi: 10.1016/S1470-2045(17)30186-9. Epub 2017 Apr 11. PMID 28410997
- [Background] Parkin DM, Stiller CA, Nectoux J. International variations in the incidence of childhood bone tumours. Int J Cancer. 1993 Feb 1;53(3):371-6. doi: 10.1002/ijc.2910530305. PMID 8428791
- [Background] Gaebler M, Silvestri A, Haybaeck J, Reichardt P, Lowery CD, Stancato LF, Zybarth G, Regenbrecht CRA. Three-Dimensional Patient-Derived In Vitro Sarcoma Models: Promising Tools for Improving Clinical Tumor Management. Front Oncol. 2017 Sep 11;7:203. doi: 10.3389/fonc.2017.00203. eCollection 2017. PMID 28955656
- [Background] Mutsaers AJ, Walkley CR. Cells of origin in osteosarcoma: mesenchymal stem cells or osteoblast committed cells? Bone. 2014 May;62:56-63. doi: 10.1016/j.bone.2014.02.003. Epub 2014 Feb 14. PMID 24530473
- [Background] Arndt CA, Crist WM. Common musculoskeletal tumors of childhood and adolescence. N Engl J Med. 1999 Jul 29;341(5):342-52. doi: 10.1056/NEJM199907293410507. No abstract available. PMID 10423470
- [Background] Howard SC, McCormick J, Pui CH, Buddington RK, Harvey RD. Preventing and Managing Toxicities of High-Dose Methotrexate. Oncologist. 2016 Dec;21(12):1471-1482. doi: 10.1634/theoncologist.2015-0164. Epub 2016 Aug 5. PMID 27496039
- [Background] Park JA, Shin HY. Influence of genetic polymorphisms in the folate pathway on toxicity after high-dose methotrexate treatment in pediatric osteosarcoma. Blood Res. 2016 Mar;51(1):50-7. doi: 10.5045/br.2016.51.1.50. Epub 2016 Mar 25. PMID 27104192
- [Background] Mazhari F, Shirazi AS, Shabzendehdar M. Management of oral mucositis in pediatric patients receiving cancer therapy: A systematic review and meta-analysis. Pediatr Blood Cancer. 2019 Mar;66(3):e27403. doi: 10.1002/pbc.27403. Epub 2018 Nov 12. PMID 30421549
- [Background] Liu SG, Gao C, Zhang RD, Zhao XX, Cui L, Li WJ, Chen ZP, Yue ZX, Zhang YY, Wu MY, Wang JX, Li ZG, Zheng HY. Polymorphisms in methotrexate transporters and their relationship to plasma methotrexate levels, toxicity of high-dose methotrexate, and outcome of pediatric acute lymphoblastic leukemia. Oncotarget. 2017 Jun 6;8(23):37761-37772. doi: 10.18632/oncotarget.17781. PMID 28525903
- [Background] Maiguma T, Hayashi Y, Ueshima S, Kaji H, Egawa T, Chayama K, Morishima T, Kitamura Y, Sendo T, Gomita Y, Teshima D. Relationship between oral mucositis and high-dose methotrexate therapy in pediatric acute lymphoblastic leukemia. Int J Clin Pharmacol Ther. 2008 Nov;46(11):584-90. doi: 10.5414/cpp46584. PMID 19000557
- [Background] Hong CHL, Gueiros LA, Fulton JS, Cheng KKF, Kandwal A, Galiti D, Fall-Dickson JM, Johansen J, Ameringer S, Kataoka T, Weikel D, Eilers J, Ranna V, Vaddi A, Lalla RV, Bossi P, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society for Oral Oncology (MASCC/ISOO). Systematic review of basic oral care for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3949-3967. doi: 10.1007/s00520-019-04848-4. Epub 2019 Jul 8. PMID 31286232
- [Background] Migliorati C, Hewson I, Lalla RV, Antunes HS, Estilo CL, Hodgson B, Lopes NN, Schubert MM, Bowen J, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of laser and other light therapy for the management of oral mucositis in cancer patients. Support Care Cancer. 2013 Jan;21(1):333-41. doi: 10.1007/s00520-012-1605-6. Epub 2012 Sep 22. PMID 23001179
- [Background] Zadik Y, Arany PR, Fregnani ER, Bossi P, Antunes HS, Bensadoun RJ, Gueiros LA, Majorana A, Nair RG, Ranna V, Tissing WJE, Vaddi A, Lubart R, Migliorati CA, Lalla RV, Cheng KKF, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of photobiomodulation for the management of oral mucositis in cancer patients and clinical practice guidelines. Support Care Cancer. 2019 Oct;27(10):3969-3983. doi: 10.1007/s00520-019-04890-2. Epub 2019 Jul 8. PMID 31286228
- [Background] He M, Zhang B, Shen N, Wu N, Sun J. A systematic review and meta-analysis of the effect of low-level laser therapy (LLLT) on chemotherapy-induced oral mucositis in pediatric and young patients. Eur J Pediatr. 2018 Jan;177(1):7-17. doi: 10.1007/s00431-017-3043-4. Epub 2017 Nov 11. PMID 29128883
- [Background] Weissheimer C, Curra M, Gregianin LJ, Daudt LE, Wagner VP, Martins MAT, Martins MD. New photobiomodulation protocol prevents oral mucositis in hematopoietic stem cell transplantation recipients-a retrospective study. Lasers Med Sci. 2017 Dec;32(9):2013-2021. doi: 10.1007/s10103-017-2314-7. Epub 2017 Aug 24. PMID 28840382
- [Background] Antunes HS, de Azevedo AM, da Silva Bouzas LF, Adao CA, Pinheiro CT, Mayhe R, Pinheiro LH, Azevedo R, D'Aiuto de Matos V, Rodrigues PC, Small IA, Zangaro RA, Ferreira CG. Low-power laser in the prevention of induced oral mucositis in bone marrow transplantation patients: a randomized trial. Blood. 2007 Mar 1;109(5):2250-5. doi: 10.1182/blood-2006-07-035022. Epub 2006 Oct 19. PMID 17053058
- [Background] Curra M, Gabriel AF, Ferreira MBC, Martins MAT, Brunetto AT, Gregianin LJ, Martins MD. Incidence and risk factors for oral mucositis in pediatric patients receiving chemotherapy. Support Care Cancer. 2021 Nov;29(11):6243-6251. doi: 10.1007/s00520-021-06199-5. Epub 2021 Apr 12. PMID 33846825
- [Background] Valer JB, Curra M, Gabriel AF, Schmidt TR, Ferreira MBC, Roesler R, Evangelista JMC, Martins MAT, Gregianin L, Martins MD. Oral mucositis in childhood cancer patients receiving high-dose methotrexate: Prevalence, relationship with other toxicities and methotrexate elimination. Int J Paediatr Dent. 2021 Mar;31(2):238-246. doi: 10.1111/ipd.12718. Epub 2020 Oct 11. PMID 32815183
- [Background] Guimaraes DM, Ota TMN, Da Silva DAC, Almeida FLDS, Schalch TD, Deana AM, Junior JMA, Fernandes KPS. Low-level laser or LED photobiomodulation on oral mucositis in pediatric patients under high doses of methotrexate: prospective, randomized, controlled trial. Support Care Cancer. 2021 Nov;29(11):6441-6447. doi: 10.1007/s00520-021-06206-9. Epub 2021 Apr 24. PMID 33893842
- [Background] Antunes HS, Herchenhorn D, Small IA, Araujo CM, Viegas CM, Cabral E, Rampini MP, Rodrigues PC, Silva TG, Ferreira EM, Dias FL, Ferreira CG. Phase III trial of low-level laser therapy to prevent oral mucositis in head and neck cancer patients treated with concurrent chemoradiation. Radiother Oncol. 2013 Nov;109(2):297-302. doi: 10.1016/j.radonc.2013.08.010. Epub 2013 Sep 14. PMID 24044799
- [Background] Sonis ST, Eilers JP, Epstein JB, LeVeque FG, Liggett WH Jr, Mulagha MT, Peterson DE, Rose AH, Schubert MM, Spijkervet FK, Wittes JP. Validation of a new scoring system for the assessment of clinical trial research of oral mucositis induced by radiation or chemotherapy. Mucositis Study Group. Cancer. 1999 May 15;85(10):2103-13. doi: 10.1002/(sici)1097-0142(19990515)85:103.0.co;2-0. PMID 10326686